CLINICAL TRIAL: NCT00835081
Title: A Two-Way , Crossover, Open-Label, Single-Dose, Fed, Bioequivalence Study of Cefadroxil 500 mg Capsules Versus DURICEF® 500 mg Capsules in Normal Healthy Non-Smoking Male and Female Subjects.
Brief Title: Cefadroxil 500 mg Capsules in Normal Healthy Non-Smoking Male and Female Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2921
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cefadroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cefadroxil 500 mg Capsules
- 2 (Active Comparator)
  Interventions: Drug: DURICEF® capsules 500 mg

INTERVENTIONS:
Drug: Cefadroxil 500 mg Capsules — 1 x 500 mg
  Arms: 1
Drug: DURICEF® capsules 500 mg — 1 x 500 mg
  Arms: 2

SUMMARY:
The objective of this study is to compare the relative bioavailability of cefadroxil 500 mg capsules (manufactured by Teva Pharmaceuticals USA) with that of DURICEF® 500 mg capsules (manufactured by Bristol-Myers Squibb Company) when dosed (1 x 500 mg capsules) in normal healthy non-smoking male and female subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female with a minimum age of 18 years (i.e. non-smoker or non-tobacco user for at least 90 days prior to pre-study medical screening.
* Body mass index (BMI= weight/height2 greater than or equal to 19kg/m2 and less than or equal to 30kg/m2.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.
* Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats/min, temperature between 35.8°C and 37.5°C.
* Negative for drugs of abuse nicotine, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum β-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides the are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria:

* Known history of hypersensitivity to cefadroxil (e.g. Duricel®) and/or related drugs in the family of cephalosporins (Cephalexin, Cefaclor, Cefazolin, Cefuroxime Axetil, Cefotetan, Cefprozil, Cefixime, Ceftriaxone), and/or penicillins (Amoxicillin, Ampicillin, Clozacillin).
* Known history or presence of fod allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of andy significant physical or organ abnormality.
* Any subject with a history of drug abuse.
* Any history or evidence of psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of over-the-counter (OTC) medication within 14 days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of contraceptives( oral, transdermal, implant, Mirena® IUD) within 30 days prior to drug administration or a depot injection or progestogen drug (e.g. Depo-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Any subject who has had blood drawn within 56 days preceding this study, during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Significant or recent history of asthma (after 12 years of age).
* Any subject with a recent(less than one year) history of alcohol abuse.
* Known personal history of gastrointestinal illness or disease, particularly colitis.
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
* Intolerance to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Tam, M.D., Principal Investigator — Biovail Contract Research
Locations (2):
- Bioassay Laboratory, Inc., Houston, Texas, United States
- Biovail Contract Research, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefadroxil (Test) First: 500 mg Cefadroxil Capsules test product dosed in first period followed by 500 mg Duricef® Capsules reference product dosed in the second period.
- Duricef® (Reference) First: 500 mg Duricef® Capsules reference product dosed in first period followed by 500 mg Cefadroxil Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Cefadroxil (Test) First | Duricef® (Reference) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Cefadroxil (Test) First | Duricef® (Reference) First
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Cefadroxil (Test) First | Duricef® (Reference) First
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefadroxil (Test) First | Duricef® (Reference) First | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 3 | 5
  Black | 3 | 3 | 6
  White | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cefadroxil (Test): 500 mg Cefadroxil Capsules test product dosed in either period.
- Duricef® (Reference): 500 mg Duricef® Capsules reference product dosed in either period.
Arm/Group | Cefadroxil (Test) | Duricef® (Reference)
Number analyzed (Participants) | 25 | 25
ng/mL | 12.024 (1.405) | 11.9 (2.688)
Statistical Analysis 1: Comparison: Cefadroxil (Test) vs Duricef® (Reference); Test type: Non-Inferiority or Equivalence — The ANOVA model containing factors for sequence of products, subjects within sequence, periods, and products was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 103, 90% CI [95.9 to 110] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefadroxil (Test) | Duricef® (Reference)
Number analyzed (Participants) | 25 | 25
ng*h/mL | 42.656 (7.063) | 42.685 (7.572)
Statistical Analysis 1: Comparison: Cefadroxil (Test) vs Duricef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100, 90% CI [97.5 to 103] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefadroxil (Test) | Duricef® (Reference)
Number analyzed (Participants) | 25 | 25
ng*h/mL | 43.987 (7.149) | 44.109 (7.631)
Statistical Analysis 1: Comparison: Cefadroxil (Test) vs Duricef® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.8, 90% CI [97.4 to 102] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.